CLINICAL TRIAL: NCT06979700
Title: Early Wake-up Predictors After Out-of-hospital Cardiac Arrest - an Observational, Multicenter Substudy of the DANOHCA Trial
Brief Title: Early WAKE-up Predictors After Out-of-Hospital Cardiac Arrest
Acronym: WAKE-OHCA
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 26745886; H-21077461 (Other: Capital Region Ethics Committee)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest (CA); Anoxic Brain Injury; Comatose Survivors of Cardiac Arrest; EEG; Pupillometry; Optic Nerve Sheath Diameter; Transcranial Doppler Ultrasound; Neurological Outcome
Keywords: wakeup; sedation
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Automated Pupillometry — Measurements will be performed on comatose participants at 0-6 hours, 20-28, 44-52 and 66-72 hours after enrolment for both pupils and include: Neurological pupil index, pupillary size, pupillary minimum diameter, pupillary constriction amplitude, pupillary constriction velocity, pupillary maximum constriction velocity, pupillary latency and pupillary dilation velocity.
Diagnostic Test: Transcranial Doppler Ultrasound — Measurements will be performed on comatose participants at 0-6 hours, 20-28, 44-52 and 66-72 hours after enrolment on both middle cerebral arteries and include the following: Peak systolic velocity, end diastolic velocity, mean velocity, pulsatility index and resistance index.
Diagnostic Test: Optic Nerve Sheath Diameter — Measurements will be performed on comatose participants at 0-6 hours, 20-28, 44-52 and 66-72 hours after enrolment on both eyes using ultrasound and include the following: optic nerve sheath diameter of right and left side and mean optic nerve sheath diameter.
Diagnostic Test: Continuous EEG and EEG Reactivity — Continuous 4-channel EEG will be established on participants as soon as possible within 0-6 hours. EEG will be stopped at successful extubation or when 72 hours has passed since study inclusion.
  EEG Reactivity will be performed on comatose participants at the following times: 0-6, 20-28, 44-52 and 66-72 hours after study inclusion. Reactivity includes 7 standardized stimuli, including 1 visual, 3 auditive and 3 pain stimuli.
  EEG data will be reviewed in Stratus EEG Analysis (Kvikna Mediacal ehf. version 5.1). Timestamps for EEG-reactivity will be manually inserted in the file. EEG Reactivity will be analysed quantitatively by power spectrum analyses performed in LabVIEW 2016 (National Instruments) according to the principles of a previous method (PMID: 36041343). Background activity within 5 minutes following reactivity stimuli, prioritizing time periods without artifacts, will be analysed by power spectrum analyses, Mindray quantitative analysis and manually analyzed by experts.

SUMMARY:
WAKE-OHCA is a prospective observational substudy of the Danish Out-of-Hospital Cardiac Arrest (DANOHCA) trial, identifier NCT05895838. The aim is to collect early neuromonitoring data to identify key predictors of successful wake-up.

DETAILED DESCRIPTION:
Background:

Post-resuscitation care following out-of-hospital cardiac arrest remains a critical area of research to optimize neurological recovery and cardiovascular outcomes. Recent findings from the Targeted Temperature Management (TTM) trials have led to the discontinuation of therapeutic hypothermia in Denmark, eliminating the need for deep sedation. The optimal sedation strategy in post-resuscitation care remains unknown, with sedation hypothesized to be neuroprotective controlling intracranial pressure but also known to be harmful and associated with adverse outcomes such as delirium, ventilator associated pneumonia, venous thromboembolism, prolonged intensive care unit (ICU) stay, delayed mobilization and patient prognostication.

Though there is emerging interest in early weaning from sedation within post-resuscitation care, limited data exist on its feasibility, prognostic implications and cost-effectiveness. Certain neuromonitoring modalities including automated pupillometry, transcranial doppler and electroencephalography (EEG) have shown promising prognostic properties, also in predicting favorable outcomes. However, sparse literature exists on early (<6 hours) prognostication related to length of sedation, and further knowledge in this area is needed to support clinical decision making.

The Danish Out-of-Hospital Cardiac Arrest (DANOHCA) study (NCT05895838) is an on-going multicenter randomized trial enrolling 1,000 participants to early wake-up (<6 hours) or standard (28-36 hours) length of sedation. This provides an opportunity to further understand neuroprognostication related to length of sedation in post-resuscitation care.

Aim and hypothesis:

This present study is designed within the context of the DANOHCA trial with the aim of identifying patient and neuromonitoring predictors of successful early and late wake-up.

The hypothesis is: Specific patient variables and neuromonitoring parameters are associated with successful wake-up.

Materials and Methods:

WAKE-OHCA will be conducted as a two-part analysis with 1) entire DANOHCA cohort (n=1,000 participants) with ICU admission data and 2) neuromonitoring data collected within the ICU on the patient cohorts at two Danish university hospital sites (Aarhus University Hospital and Rigshospitalet) during the study inclusion period (anticipated n=250 participants, with the exception of n=100 participants for EEG measurements, as these will only be performed at Aarhus University Hospital site).

DANOHCA inclusion criteria are: Out-of-hospital cardiac arrest of a presumed cardiac cause, age > 18 years, sustained return of spontaneous circulation for more than 20 minutes, unconscious upon admission.

The first part will include baseline characteristics, cardiac arrest data, and initial biochemistry. Data is collected from Danish prehospital patient journal (PPJ), electronic patient journals (EPJ, Sundhedsplatformen), Danish cardiac arrest registry and DANOHCA patient database.

The second part will include the following non-invasive neuromonitoring data collected prospectively at 0-6 hours, 20-28 hours, 44-52 hours and 66-72 hours after enrolment:

* Bilateral automated pupillometry
* Transcranial doppler evaluating both middle cerebral arteries.
* Bilateral Optic Nerve Sheath Diameter measured by ultrasound.
* Continuous 4-channel EEG background activity and EEG reactivity tests.

These will provide insight on early neurological status and recovery patterns, cerebral hemodynamics and intracranial pressure. Neuromonitoring data will only be collected on participants that are still comatose. Clinicians will be blinded from collected data, and it will have no impact on participants' treatment.

Automated pupillometry will be done with a NeurOptics NPi-200 pupillometer (NeurOptics, Irvine, California, USA). Transcranial doppler and ONSD measurements will be conducted with a Vivid S70N (GE Healthcare, Chicago, IL, USA) and analysed using Echopac (GE Healthcare, Chicago, IL, USA). EEG measurements will be done with Mindray BeneVision N-series with an aEEG module (Shenzhen Mindray Bio-Medical Electronics Co., Nanshan, Shenzhen, China).

Logistic regression analysis will be conducted to explore the association between participant and neuromonitoring variables and successful wake-up with unsuccessful wake-up as reference group. Secondary analyses will investigate how neuromonitoring variables perform in predicting patient outcomes (mortality, neurological outcome) in the early and late wake-up groups as well as how serial neuromonitoring variables are associated with successful wake-up at later stages.

Significance:

By identifying key predictors of early wake-up success, this project may refine patient selection, optimize individualized treatment, and enhance prognostication. Insights into neuromonitoring could improve clinical decision-making and reduce unnecessary sedation, minimizing associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* OHCA of presumed cardiac cause
* Sustained ROSC, defined as persistent signs of circulation and no need for chest compressions or mechanical circulatory support for 20 minutes
* Unconsciousness (GCS <9) (patients not able to obey verbal commands) after sustained ROSC at the time of randomization

Exclusion Criteria:

* Females of childbearing potential if pregnancy is suspected (unless a negative HCG test can rule out pregnancy within the inclusion window)
* Known bleeding diathesis (medically induced coagulopathy (e.g. warfarin, NOAC, clopidogrel) does not exclude the patient)
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Unwitnessed asystole
* Known limitations in therapy and Do Not Resuscitate-order
* Known disease making 180 days survival unlikely
* Known pre-arrest CPC 3 or 4 functional status
* >3 hours (180 minutes) from ROSC to screening
* Systolic blood pressure <80 mm Hg despite fluid loading/vasopressor and/or inotropic medication (If the systolic blood pressure is recovering during the inclusion window of 180 minutes the patient may be included)
* Use of intra-aortic balloon pump/axial flow device/ECMO (If the patient is weaned and the device is removed during the inclusion window of 180 minutes the patient may be included)
* Temperature on admission <30°C
* Known allergy for dexamethasone or olanzapine
* Ongoing (within 48 h) treatment with olanzapine or dexamethasone
* Known back or hip condition that precluded the patients from being positioned with backrest from 0 to 45-degree angle
* Known or suspected Long QT Syndrome (LQTS)
* Known active fungal disease. Localized skin lesions do not exclude patients from inclusion
* Estimated body weight <45kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the DANOHCA trial at Aarhus University Hospital and Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful wake-up | 0-6 hours or 28-36 hours according to DANOHCA randomization.
  Defined as awake and successfully extubated.

SECONDARY OUTCOMES:
Number of patients with successful delayed wake-up | Up to 90 days.
  Defined as awake and successfully extubated later than according to DANOHCA randomization.
Duration of intubation | Up to 90 days.
  Assessed as the duration of intubation from randomization till extubation during initial ICU stay (oral and tracheostomy combined).
Days alive outside hospital | 30 days.
  Counted as days alive outside of hospital after discharge.
30-day mortality | 30 days.
  Number of patients dying from all causes.
90-day mortality | 90 days.
  Number of patients dying from all causes.
Length of ICU stay | From randomization till discharge from the ICU, up to 90 days.
  Assessed as the initial ICU length of stay.
Length of hospital stay | From randomization till discharge from hospital or in-patient rehabilitation, up to 90 days.
  Assessed as the hospital length of stay (including in-patient rehabilitation and transfer to referral hospital).
Cerebral Performance Category (CPC) | Up to 6 months.
  CPC score at ICU discharge, at hospital discharge, and at ambulatory follow-up (scheduled visit at 3 to 6 months after the cardiac arrest). The CPC score ranges from 1 to 5 with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD, DMSc, Study Chair — Department of Cardiology, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Intensive Care Medicine, Aarhus N
  - Department of Cardiology, The Heart Centre, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No